CLINICAL TRIAL: NCT02460224
Title: A Phase I/II, Open Label, Multicenter Study of the Safety and Efficacy of LAG525 Single Agent and in Combination With PDR001 Administered to Patients With Advanced Malignancies
Brief Title: Safety and Efficacy of LAG525 Single Agent and in Combination With PDR001 in Patients With Advanced Malignancies.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAG525X2101C; 2015-000449-21 (EudraCT Number)
Record Dates: First submitted 2015-05-09; First posted 2015-06-02 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors
Keywords: Non-small cell lung cancer; Melanoma; Renal cancer; Mesothelioma; Triple Negative Breast; TNBC; Renal
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Kidney Neoplasms; Mesothelioma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (29):
- Phase 1: LAG525 1 mg/kg Q2W (Experimental): Single-agent LAG525 1 mg/kg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 3 mg/kg Q2W (Experimental): Single-agent LAG525 3 mg/kg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 5 mg/kg Q2W (Experimental): Single-agent LAG525 5 mg/kg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 10 mg/kg Q2W (Experimental): Single-agent LAG525 10 mg/kg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 15 mg/kg Q2W (Experimental): Single-agent LAG525 15 mg/kg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 240 mg Q2W (Experimental): Single-agent LAG525 240 mg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 400 mg Q2W (Experimental): Single-agent LAG525 400 mg Q2W
  Interventions: Drug: LAG525
- Phase 1: LAG525 3 mg/kg Q4W (Experimental): Single-agent LAG525 3 mg/kg Q4W
  Interventions: Drug: LAG525
- Phase 1: LAG525 5 mg/kg Q4W (Experimental): Single-agent LAG525 5 mg/kg Q4W
  Interventions: Drug: LAG525
- Phase 1: LAG525 10 mg/kg Q4W (Experimental): Single-agent LAG525 10 mg/kg Q4W
  Interventions: Drug: LAG525
- Phase 1: LAG525 400 mg Q4W (Experimental): Single-agent LAG525 400 mg Q4W
  Interventions: Drug: LAG525
- Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W (Experimental): Combination LAG525 0.3 mg/kg + PDR001 1 mg/kg (Q2W/Q2W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W (Experimental): Combination LAG525 1 mg/kg + PDR001 1 mg/kg (Q2W/Q2W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W (Experimental): Combination LAG525 80 mg + PDR001 80 mg (Q2W/Q2W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W (Experimental): Combination LAG525 80 mg + PDR001 240 mg (Q2W/Q2W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W (Experimental): Combination LAG525 240 mg + PDR001 240 mg (Q2W/Q2W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W (Experimental): Combination LAG525 240 mg + PDR001 300 mg (Q3W/Q3W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W (Experimental): Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W (Experimental): Combination LAG525 600 mg + PDR001 300 mg (Q3W/Q3W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W (Experimental): Combination LAG525 80 mg + PDR001 240 mg (Q4W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W (Experimental): Combination LAG525 400 mg + PDR001 400 mg (Q4W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W (Experimental): Combination LAG525 800 mg + PDR001 400 mg (Q4W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W (Experimental): Combination LAG525 1000 mg + PDR001 400 mg (Q4W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W (Experimental): Combination LAG525 80 mg + PDR001 400 mg (Q2W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W (Experimental): Combination LAG525 240 mg + PDR001 400 mg (Q2W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W (Experimental): Combination LAG525 300 mg + PDR001 400 mg (Q2W/Q4W)
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W (Experimental): Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients naïve to anti-PD-1/PD-L1
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W (Experimental): Combination LAG525 600 mg + PDR001 400 mg (Q4W/Q4W) in patients naïve to anti-PD-1/PD-L1
  Interventions: Drug: LAG525; Drug: PDR001
- Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W (Experimental): Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients pre-treated with anti-PD-1/PD-L1
  Interventions: Drug: LAG525; Drug: PDR001

INTERVENTIONS:
Drug: LAG525 — LAG525 was administered via intravenous (i.v.) infusion
Drug: PDR001 — PDR001 was administered via i.v. infusion
  Arms: Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W; Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W; Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W; Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W; Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W; Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W; Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W; Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W; Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W; Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W; Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W; Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W; Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W; Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W; Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W; Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W; Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W; Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W

SUMMARY:
This study was to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of LAG525 as a single agent and in combination with PDR001 to adult patients with solid tumors. The study consists of a dose escalation (phase 1) to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) for LAG525 as a single agent and in combination with PDR001, and a dose expansion (phase 2) which characterized treatment of LAG525 in combination with PDR001 at the MTD or RP2D.

DETAILED DESCRIPTION:
This was a Phase 1/2, multi-center, open-label study comprising a Phase 1 dose escalation part followed by a Phase 2 dose expansion part.

During the Phase 1 dose escalation part patients with any advanced solid tumor received the study treatment until the MTD was reached or a lower RP2D was established. The study had the following 3 dose escalation parts: 1) Single-agent LAG525; 2) Single-agent LAG525 in Japanese patients; 3) Combination of LAG525 with PDR001.

Once the RP2D or MTD had been determined in the escalation parts, additional patients were to be enrolled in the Phase 2 expansion parts in order to assess the preliminary anti-tumor activity. Phase 2 expansion cohorts testing single-agent LAG525 were not opened for enrollment based on emerging data including but not limited to preliminary anti-tumor activity. Phase 2 expansion cohorts for the combination of LAG525 with PDR001 were opened and 5 tumor types were assessed: 1) Non-small cell lung cancer (NSCLC); 2) Melanoma; 3) Renal cell cancer (RCC); 4) Mesothelioma; 5) Triple negative breast cancer (TNBC). The efficacy and safety of the combination of LAG525 with PDR001 in these tumor types was assessed in both the PD-1/PD-L1 pre-treated and naïve settings.

ELIGIBILITY:
Inclusion Criteria:

Phase I part:

- Patients with advanced/metastatic solid tumors, with measurable or non-measurable disease as determined by RECIST version 1.1, who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists

Phase II part:

* Patients with advanced/metastatic solid tumors, with at least one measurable lesion as determined by RECIST version 1.1, who have had disease progression following their last prior therapy and fit into one of the following groups:
* Group 1: NSCLC
* Group 2: Melanoma
* Group 3: Renal cancer
* Group 4: Mesothelioma
* Group 5: TNBC
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Patient must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy.

Exclusion Criteria:

* History of severe hypersensitivity reactions to study treatment ingredients or other mAbs
* Active, known or suspected autoimmune disease
* Active infection requiring systemic antibiotic therapy
* HIV infection. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Patients receiving chronic treatment with systemic steroid therapy, other than replacement-dose corticosteroids in the setting of adrenal insufficiency
* Patients receiving systemic treatment with any immunosuppressive medication
* Use of live vaccines against infectious disease within 4 weeks of initiation of study treatment
* Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment.
* Presence of symptomatic central nervous system (CNS) metastases or CNS metastases that require local CNS-directed therapy or increasing doses of corticosteroids within the prior 2 weeks
* History of drug-induced pneumonitis or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (6):
  - Columbia University Medical Center SC LAG X2101C, New York, New York
  - Memorial Sloan Kettering Cancer Center SC, New York, New York
  - Duke Clinical Research Institute SC, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center UT Health Science Center CTRC 2, San Antonio, Texas
  - Huntsman Cancer Institute Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria
- Novartis Investigative Site, Leuven, Belgium
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Toronto, Ontario
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Saint-Herblain Cédex
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Fukuoka, Fukuoka, Japan
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rivoltini L, Camisaschi C, Fuca G, Paolini B, Vergani B, Beretta V, Damian S, Duca M, Cresta S, Magni M, Leone BE, Castelli C, de Braud F, De Santis F, Di Nicola M. Immunological characterization of a long-lasting response in a patient with metastatic triple-negative breast cancer treated with PD-1 and LAG-3 blockade. Sci Rep. 2024 Feb 9;14(1):3379. doi: 10.1038/s41598-024-54041-9. PMID 38336861
- [Derived] Schoffski P, Tan DSW, Martin M, Ochoa-de-Olza M, Sarantopoulos J, Carvajal RD, Kyi C, Esaki T, Prawira A, Akerley W, De Braud F, Hui R, Zhang T, Soo RA, Maur M, Weickhardt A, Krauss J, Deschler-Baier B, Lau A, Samant TS, Longmire T, Chowdhury NR, Sabatos-Peyton CA, Patel N, Ramesh R, Hu T, Carion A, Gusenleitner D, Yerramilli-Rao P, Askoxylakis V, Kwak EL, Hong DS. Phase I/II study of the LAG-3 inhibitor ieramilimab (LAG525) +/- anti-PD-1 spartalizumab (PDR001) in patients with advanced malignancies. J Immunother Cancer. 2022 Feb;10(2):e003776. doi: 10.1136/jitc-2021-003776. PMID 35217575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 25 investigative sites in 12 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. All screening/baseline evaluations were performed ≤ 21 days before Cycle 1 Day 1, except for baseline radiological evaluations which had to be done within 28 days.
Period: Overall Study
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Started | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6 | 121 | 21 | 93
Rest of the World Patients in the Dose Escalation Part | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6 | 0 | 0 | 0
Japanese Patients in the Dose Escalation Part | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6 | 121 | 21 | 93
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 11 | 1 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 14 | 1 | 6
Not completed — Progressive disease | 15 | 11 | 5 | 6 | 3 | 26 | 28 | 4 | 5 | 9 | 5 | 4 | 5 | 4 | 5 | 5 | 15 | 3 | 8 | 3 | 4 | 9 | 4 | 11 | 4 | 5 | 85 | 17 | 77
Not completed — Subject/guardian decision | 2 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Total
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6 | 121 | 21 | 93 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.55) | 64.5 (12.43) | 61.8 (13.32) | 53.3 (20.76) | 61.2 (9.58) | 57.2 (10.94) | 56.7 (10.82) | 60.8 (9.36) | 54.8 (17.26) | 59.5 (7.16) | 60.4 (7.16) | 54.3 (8.78) | 58.0 (5.90) | 44.8 (5.23) | 58.2 (10.03) | 48.7 (24.36) | 59.1 (12.83) | 61.2 (11.34) | 61.3 (8.25) | 51.1 (12.03) | 59.8 (8.11) | 51.8 (12.10) | 59.2 (5.42) | 56.6 (10.31) | 60.7 (6.89) | 52.3 (12.50) | 61.0 (10.79) | 49.4 (8.94) | 58.4 (11.18) | 58.1 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 3 | 4 | 4 | 17 | 14 | 2 | 4 | 6 | 2 | 3 | 3 | 2 | 1 | 3 | 9 | 3 | 11 | 3 | 3 | 7 | 5 | 6 | 4 | 3 | 53 | 20 | 40 | 248
  Male | 10 | 6 | 3 | 2 | 2 | 13 | 16 | 3 | 2 | 5 | 3 | 3 | 3 | 4 | 4 | 3 | 11 | 3 | 1 | 4 | 3 | 5 | 1 | 5 | 2 | 3 | 68 | 1 | 53 | 242
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 9 | 5 | 3 | 6 | 20 | 20 | 2 | 4 | 10 | 3 | 2 | 6 | 6 | 4 | 5 | 20 | 6 | 10 | 7 | 4 | 8 | 5 | 9 | 5 | 6 | 69 | 15 | 70 | 347
  Black | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
  Asian | 8 | 2 | 1 | 3 | 0 | 10 | 10 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 2 | 1 | 0 | 48 | 4 | 17 | 122
  Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 12
  Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment with single-agent LAG525 or within the first two cycles of treatment with the combination of LAG525 and PDR001. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Time Frame: 15 days for single-agent LAG525 arms and 30 days for the combination LAG525 + PDR001 arms
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001, and who either completed a minimum exposure requirement or who had a DLT during the first 15 days of treatment (1 cycle) for single-agent LAG525 arms or the first 30 days (2 cycles) for the LAG525 + PDR001 arms.
  Japanese patients were analyzed together with the rest of the world (ROW) patients as per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 16 | 12 | 6 | 5 | 6 | 28 | 27 | 5 | 6 | 11 | 5 | 6 | 6 | 5 | 5 | 5 | 17 | 4 | 9 | 5 | 6 | 11 | 6 | 11 | 5 | 6
Participants | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0

2. Primary Outcome: Phase 2: Overall Response Rate (ORR) Per RECIST 1.1
Description: Tumor response was based on local investigator assessment and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). ORR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
  ORR is reported by tumor type.
Time Frame: From start of treatment until end of treatment, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
percentage of participants
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  Non-small cell lung cancer (NSCLC) | 15.0 [4.2 to 34.4] |  | 0 [0.0 to 12.7]
  Melanoma: number analyzed (Participants) | 20 | 0 | 22
  Melanoma | 15.0 [4.2 to 34.4] |  | 9.1 [1.6 to 25.9]
  Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  Renal cell cancer (RCC) | 26.3 [11.0 to 47.6] |  | 5.3 [0.3 to 22.6]
  Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  Mesothelioma | 17.1 [8.3 to 29.7] |  | 6.3 [0.3 to 26.4]
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  Triple negative breast cancer (TNBC) | 14.3 [4.0 to 32.9] | 4.8 [0.2 to 20.7] | 0 [0.0 to 19.3]

3. Secondary Outcome: Phase 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs. The number of participants in each category (Rest of the World (ROW) patients, Japanese patients) with AEs and SAEs are reported in this record.
Time Frame: From first dose of study treatment until last dose of study treatment plus 30 days post treatment, assessed up to 4.5 years.
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
Participants
  AEs, ROW patients: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  AEs, ROW patients | 13 | 11 | 6 | 6 | 6 | 24 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 19 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  SAEs, ROW patients: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  SAEs, ROW patients | 4 | 2 | 5 | 2 | 3 | 10 | 11 | 2 | 4 | 5 | 2 | 3 | 2 | 3 | 3 | 1 | 9 | 3 | 6 | 4 | 5 | 5 | 2 | 5 | 4 | 4
  AEs, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs, Japanese patients | 4 |  |  |  |  | 5 | 6 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  SAEs, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAEs, Japanese patients | 0 |  |  |  |  | 2 | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

4. Secondary Outcome: Phase 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs. The number of participants with AEs and SAEs is reported for each tumor type.
Time Frame: From first dose of study treatment until last dose of study treatment plus 30 days post treatment, assessed up to 2.7 years.
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
Participants
  AEs, Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  AEs, Non-small cell lung cancer (NSCLC) | 19 |  | 22
  SAEs, Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  SAEs, Non-small cell lung cancer (NSCLC) | 13 |  | 7
  AEs, Melanoma: number analyzed (Participants) | 20 | 0 | 22
  AEs, Melanoma | 19 |  | 22
  SAEs, Melanoma: number analyzed (Participants) | 20 | 0 | 22
  SAEs, Melanoma | 8 |  | 8
  AEs, Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  AEs, Renal cell cancer (RCC) | 19 |  | 19
  SAEs, Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  SAEs, Renal cell cancer (RCC) | 14 |  | 5
  AEs, Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  AEs, Mesothelioma | 41 |  | 16
  SAEs, Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  SAEs, Mesothelioma | 15 |  | 4
  AEs, Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  AEs, Triple negative breast cancer (TNBC) | 21 | 21 | 14
  SAEs, Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  SAEs, Triple negative breast cancer (TNBC) | 9 | 10 | 4

5. Secondary Outcome: Phase 1: Number of Participants With Dose Reductions and Dose Interruptions of LAG525 and PDR001
Description: Number of participants with at least one dose reduction of LAG525, at least one dose interruption of LAG525, at least one dose reduction of PDR001 and at least one dose interruption of PDR001.
  Japanese patients were not treated with PDR001 and therefore the dose reductions and dose interruptions of this study drug are not applicable.
Time Frame: From start of treatment until end of treatment, assessed up to 4.4 years.
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
Participants
  LAG525 dose reduction, ROW patients: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  LAG525 dose reduction, ROW patients | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  LAG525 dose interruption, ROW patients: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  LAG525 dose interruption, ROW patients | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 4 | 1 | 2 | 1 | 1 | 6 | 2 | 2 | 1 | 2 | 3 | 0 | 4 | 1 | 1
  PDR001 dose reduction, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  PDR001 dose reduction, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  PDR001 dose interruption, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  PDR001 dose interruption, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 4 | 1 | 2 | 1 | 0 | 6 | 2 | 2 | 1 | 2 | 3 | 0 | 3 | 0 | 1
  LAG525 dose reduction, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LAG525 dose reduction, Japanese patients | 0 |  |  |  |  | 0 | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  LAG525 dose interruption, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LAG525 dose interruption, Japanese patients | 0 |  |  |  |  | 2 | 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

6. Secondary Outcome: Phase 2: Number of Participants With Dose Reductions and Dose Interruptions of LAG525 and PDR001
Description: Number of participants with at least one dose reduction of LAG525, at least one dose interruption of LAG525, at least one dose reduction of PDR001 and at least one dose interruption of PDR001.
  The number of participants with dose reductions and dose interruptions of both study drugs is reported for each tumor type.
Time Frame: From start of treatment until end of treatment, assessed up to 2.6 years.
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
Participants
  LAG525 dose reduction, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  LAG525 dose reduction, NSCLC patients | 0 |  | 0
  LAG525 dose interruption, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  LAG525 dose interruption, NSCLC patients | 3 |  | 3
  PDR001 dose reduction, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  PDR001 dose reduction, NSCLC patients | 0 |  | 0
  PDR001 dose interruption, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  PDR001 dose interruption, NSCLC patients | 3 |  | 3
  LAG525 dose reduction, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  LAG525 dose reduction, melanoma patients | 0 |  | 0
  LAG525 dose interruption, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  LAG525 dose interruption, melanoma patients | 4 |  | 4
  PDR001 dose reduction, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  PDR001 dose reduction, melanoma patients | 0 |  | 0
  PDR001 dose interruption, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  PDR001 dose interruption, melanoma patients | 4 |  | 4
  LAG525 dose reduction, RCC patients: number analyzed (Participants) | 19 | 0 | 19
  LAG525 dose reduction, RCC patients | 0 |  | 0
  LAG525 dose interruption, RCC patients: number analyzed (Participants) | 19 | 0 | 19
  LAG525 dose interruption, RCC patients | 5 |  | 1
  PDR001 dose reduction, RCC patients: number analyzed (Participants) | 19 | 0 | 19
  PDR001 dose reduction, RCC patients | 0 |  | 0
  PDR001 dose interruption, RCC patients: number analyzed (Participants) | 19 | 0 | 19
  PDR001 dose interruption, RCC patients | 5 |  | 1
  LAG525 dose reduction, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  LAG525 dose reduction, mesothelioma patients | 0 |  | 0
  LAG525 dose interruption, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  LAG525 dose interruption, mesothelioma patients | 8 |  | 5
  PDR001 dose reduction, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  PDR001 dose reduction, mesothelioma patients | 0 |  | 0
  PDR001 dose interruption, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  PDR001 dose interruption, mesothelioma patients | 8 |  | 5
  LAG525 dose reduction, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  LAG525 dose reduction, TNBC patients | 0 | 0 | 0
  LAG525 dose interruption, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  LAG525 dose interruption, TNBC patients | 3 | 0 | 0
  PDR001 dose reduction, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  PDR001 dose reduction, TNBC patients | 0 | 0 | 0
  PDR001 dose interruption, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  PDR001 dose interruption, TNBC patients | 3 | 0 | 0

7. Secondary Outcome: Phase 1: Relative Dose Intensity (RDI) of LAG525 and PDR001
Description: Relative dose intensity of each study drug is calculated with the following formula: 100 x actual dose intensity (mg/day)/planned dose intensity (mg/day).
  Japanese patients were not treated with PDR001 and therefore the RDI of this study drug is not applicable.
Time Frame: From start of treatment until end of treatment, assessed up to 4.4 years.
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
percentage
  LAG525, ROW patients: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  LAG525, ROW patients | 98.9 (3.93) | 100 (0) | 94.4 (13.61) | 100 (0) | 98.2 (4.47) | 99.0 (5.00) | 99.9 (0.60) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 97.4 (6.27) | 100 (0) | 99.7 (0.84) | 100 (0) | 99.6 (0.93) | 97.8 (5.27) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 97.7 (7.54) | 100 (0) | 100 (0)
  PDR001, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  PDR001, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 97.3 (6.72) | 100 (0) | 97.6 (5.00) | 100 (0) | 100 (0) | 98.0 (4.95) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0) | 100 (0)
  LAG525, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LAG525, Japanese patients | 100 (0) |  |  |  |  | 98.0 (4.47) | 100 (0) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

8. Secondary Outcome: Phase 2: Relative Dose Intensity (RDI) of LAG525 and PDR001
Description: Relative dose intensity of each study drug is calculated with the following formula: 100 x actual dose intensity (mg/day)/planned dose intensity (mg/day).
  The RDI of both study drugs is reported for each tumor type.
Time Frame: From start of treatment until end of treatment, assessed up to 2.6 years.
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
percentage
  LAG525, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  LAG525, NSCLC patients | 100 (0) |  | 100 (0)
  PDR001, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  PDR001, NSCLC patients | 100 (0) |  | 99.8 (0.71)
  LAG525, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  LAG525, melanoma patients | 99.4 (2.80) |  | 99.7 (1.47)
  PDR001, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  PDR001, melanoma patients | 99.4 (2.80) |  | 99.7 (1.47)
  LAG525, RCC patients: number analyzed (Participants) | 19 | 0 | 19
  LAG525, RCC patients | 100 (0) |  | 100 (0)
  PDR001, RCC patients: number analyzed (Participants) | 19 | 0 | 19
  PDR001, RCC patients | 100 (0) |  | 100 (0)
  LAG525, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  LAG525, mesothelioma patients | 99.3 (4.26) |  | 99.4 (1.99)
  PDR001, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  PDR001, mesothelioma patients | 99.3 (4.26) |  | 99.4 (1.99)
  LAG525, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  LAG525, TNBC patients | 96.5 (11.08) | 100 (0) | 100 (0)
  PDR001, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  PDR001, TNBC patients | 98.4 (7.21) | 100 (0) | 100 (0)

9. Secondary Outcome: Phase 1: Maximum Observed Serum Concentration (Cmax) of LAG525
Description: Pharmacokinetic (PK) parameters were calculated based on LAG525 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-infusion, 1, 24, 168, 240 and 336 hours post-infusion, and 504 hours (Q3W regimens only) and 672 hours (Q4W regimens only) post infusion on Cycle 1 Day 1 and Cycle 3 Day 1. The duration of one cycle was 14 days (Q2W), 21 days (Q3W) and 28 days (Q4W).
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 and who had at least one serum sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 29 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
ug/mL
  Cycle 1, ROW patients: number analyzed (Participants) | 12 | 12 | 6 | 6 | 6 | 24 | 23 | 5 | 6 | 6 | 5 | 6 | 5 | 6 | 4 | 6 | 16 | 3 | 9 | 7 | 3 | 9 | 5 | 9 | 5 | 6
  Cycle 1, ROW patients | 21.8 (6.52) | 72.4 (14.1) | 117 (26.7) | 247 (63.2) | 393 (95.2) | 73.8 (19.2) | 116 (28.3) | 66.4 (14.1) | 118 (23.8) | 268 (38.5) | 125 (38.9) | 8.58 (2.53) | 26.5 (3.6) | 24.1 (6.58) | 25.1 (6.81) | 87.9 (24.7) | 73.1 (14.7) | 122 (36.4) | 215 (43.9) | 27.2 (5.51) | 121 (8.96) | 276 (66.5) | 303 (82.3) | 27.1 (7.56) | 86.2 (22.2) | 73.1 (42.2)
  Cycle 3, ROW patients: number analyzed (Participants) | 4 | 7 | 1 | 1 | 3 | 9 | 9 | 3 | 2 | 2 | 2 | 3 | 4 | 3 | 3 | 4 | 14 | 2 | 5 | 3 | 2 | 4 | 2 | 6 | 5 | 3
  Cycle 3, ROW patients | 34.7 (13.2) | 124 (30.5) | 272 | 306 | 607 (108) | 114 (36.5) | 169 (60.7) | 77.9 (11) | 117 (26.2) | 222 (0) | 250 (187) | 9.57 (4.91) | 31.6 (9.9) | 35.2 (7.29) | 33.8 (7.75) | 156 (70.4) | 88.7 (25.3) | 114 (19.8) | 274 (57.1) | 32 (17) | 174 (11.3) | 354 (118) | 513 (72.8) | 33.3 (14.5) | 96 (42.8) | 147 (43)
  Cycle 1, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Japanese patients | 23.1 (2.58) |  |  |  |  | 95.5 (18.3) | 152 (33.9) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3, Japanese patients: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3, Japanese patients | 32.6 (1.2) |  |  |  |  | 198 | 255 (59.1) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

10. Secondary Outcome: Phase 2: Maximum Observed Serum Concentration (Cmax) of LAG525
Description: as for outcome 9
Time Frame: pre-infusion, 1, 24, 168, 240 and 336 hours post-infusion, and 504 hours (Q3W regimens only) and 672 hours (Q4W regimens only) post infusion on Cycle 1 Day 1 and Cycle 3 Day 1. The duration of one cycle was 21 days (Q3W) and 28 days (Q4W).
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 and who had at least one serum sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 92
ug/mL
  Cycle 1, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  Cycle 1, NSCLC patients | 154 (43.5) |  | 106 (26.8)
  Cycle 3, NSCLC patients: number analyzed (Participants) | 15 | 0 | 15
  Cycle 3, NSCLC patients | 169 (51.9) |  | 137 (30.8)
  Cycle 1, melanoma patients: number analyzed (Participants) | 20 | 0 | 21
  Cycle 1, melanoma patients | 115 (29.9) |  | 102 (36.7)
  Cycle 3, melanoma patients: number analyzed (Participants) | 13 | 0 | 14
  Cycle 3, melanoma patients | 171 (32) |  | 163 (52.8)
  Cycle 1, RCC patients: number analyzed (Participants) | 18 | 0 | 16
  Cycle 1, RCC patients | 118 (34.7) |  | 111 (28.3)
  Cycle 3, RCC patients: number analyzed (Participants) | 13 | 0 | 11
  Cycle 3, RCC patients | 158 (45.4) |  | 153 (43.5)
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 40 | 0 | 15
  Cycle 1, mesothelioma patients | 116 (31) |  | 119 (37.6)
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 32 | 0 | 15
  Cycle 3, mesothelioma patients | 141 (39.7) |  | 138 (33.1)
  Cycle 1, TNBC patients: number analyzed (Participants) | 21 | 21 | 13
  Cycle 1, TNBC patients | 144 (32.4) | 207 (53.1) | 132 (26.7)
  Cycle 3, TNBC patients: number analyzed (Participants) | 10 | 4 | 9
  Cycle 3, TNBC patients | 179 (65.2) | 190 (55) | 157 (33.2)

11. Secondary Outcome: Phase 1: Time to Reach Maximum Serum Concentration (Tmax) of LAG525
Description: Pharmacokinetic (PK) parameters were calculated based on LAG525 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 29 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
days
  Cycle 1, ROW patients: number analyzed (Participants) | 12 | 12 | 6 | 6 | 6 | 24 | 23 | 5 | 6 | 6 | 5 | 6 | 5 | 6 | 4 | 6 | 16 | 3 | 9 | 7 | 3 | 9 | 5 | 9 | 5 | 6
  Cycle 1, ROW patients | 1.73 [1.5 to 2.45] | 1.6 [1.1 to 2.62] | 1.63 [1.17 to 2.13] | 1.63 [1.5 to 2.35] | 1.99 [1.48 to 2.07] | 1.59 [1.5 to 2.17] | 1.57 [1.47 to 2.45] | 1.58 [1.03 to 2.25] | 2.1 [1.5 to 2.17] | 2.02 [1.5 to 2.28] | 1.5 [1.5 to 1.68] | 1.5 [1.5 to 1.65] | 1.5 [0.933 to 1.53] | 1.5 [1.47 to 1.52] | 1.53 [1.5 to 1.58] | 1.55 [1.5 to 2.03] | 1.52 [1.02 to 4.25] | 1.5 [1.5 to 1.58] | 1.57 [1 to 4.45] | 1.52 [1.5 to 1.55] | 1.5 [1.5 to 1.5] | 1.58 [1.5 to 2.07] | 1.58 [1.5 to 2.1] | 1.5 [1.5 to 2.57] | 1.7 [1.57 to 2.08] | 1.5 [0 to 1.55]
  Cycle 3, ROW patients: number analyzed (Participants) | 4 | 7 | 1 | 1 | 3 | 9 | 9 | 3 | 2 | 2 | 2 | 3 | 4 | 3 | 3 | 4 | 14 | 2 | 5 | 3 | 2 | 4 | 2 | 6 | 5 | 3
  Cycle 3, ROW patients | 1.83 [1.5 to 2.12] | 2.05 [1.55 to 2.08] | 1.08 [1.08 to 1.08] | 1.55 [1.55 to 1.55] | 1.67 [1.67 to 2.08] | 1.58 [1.33 to 2.05] | 1.5 [1.5 to 2.55] | 2.08 [1.52 to 2.12] | 1.93 [1.57 to 2.3] | 1.83 [1.65 to 2] | 1.5 [1.5 to 1.5] | 1.72 [1.57 to 1.83] | 1.51 [1.5 to 1.57] | 1.5 [1.5 to 1.58] | 1.5 [1.5 to 1.52] | 1.53 [1.5 to 2] | 1.53 [1.48 to 3.77] | 1.58 [1.58 to 1.58] | 1.52 [1 to 1.55] | 1.58 [1.5 to 1.75] | 1.54 [1.5 to 1.58] | 1.58 [1.5 to 2.05] | 1.75 [1.5 to 2] | 1.53 [1.5 to 2.55] | 1.58 [0 to 2] | 1.58 [1.57 to 1.58]
  Cycle 1, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Japanese patients | 1.58 [1.55 to 1.68] |  |  |  |  | 1.54 [1.5 to 1.63] | 1.54 [1.52 to 1.55] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3, Japanese patients: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3, Japanese patients | 1.63 [1.58 to 1.68] |  |  |  |  | 1.57 [1.57 to 1.57] | 1.6 [1.55 to 1.67] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

12. Secondary Outcome: Phase 2: Time to Reach Maximum Serum Concentration (Tmax) of LAG525
Description: as for outcome 11
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: days
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 92
days
  Cycle 1, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  Cycle 1, NSCLC patients | 1.53 [0.917 to 3] |  | 1.55 [0.917 to 2.62]
  Cycle 3, NSCLC patients: number analyzed (Participants) | 15 | 0 | 15
  Cycle 3, NSCLC patients | 1.55 [1.45 to 2] |  | 1.58 [1.5 to 2.33]
  Cycle 1, melanoma patients: number analyzed (Participants) | 20 | 0 | 21
  Cycle 1, melanoma patients | 1.51 [1.43 to 3] |  | 1.53 [1.07 to 2.9]
  Cycle 3, melanoma patients: number analyzed (Participants) | 13 | 0 | 14
  Cycle 3, melanoma patients | 1.53 [1.45 to 2] |  | 1.53 [0.683 to 1.82]
  Cycle 1, RCC patients: number analyzed (Participants) | 18 | 0 | 16
  Cycle 1, RCC patients | 1.51 [1 to 3] |  | 1.53 [1 to 2.05]
  Cycle 3, RCC patients: number analyzed (Participants) | 13 | 0 | 11
  Cycle 3, RCC patients | 1.58 [1.48 to 2.08] |  | 1.53 [1.45 to 2.8]
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 40 | 0 | 15
  Cycle 1, mesothelioma patients | 1.53 [0.583 to 3] |  | 1.55 [1.47 to 2.08]
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 32 | 0 | 15
  Cycle 3, mesothelioma patients | 1.5 [0.967 to 2.13] |  | 1.52 [1.42 to 2.08]
  Cycle 1, TNBC patients: number analyzed (Participants) | 21 | 21 | 13
  Cycle 1, TNBC patients | 1.53 [0.567 to 3] | 1.53 [1.43 to 3] | 1.58 [0.95 to 2]
  Cycle 3, TNBC patients: number analyzed (Participants) | 10 | 4 | 9
  Cycle 3, TNBC patients | 1.63 [1.48 to 2] | 1.78 [1.7 to 1.92] | 1.6 [1 to 2]

13. Secondary Outcome: Phase 1: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of LAG525
Description: Pharmacokinetic (PK) parameters were calculated based on LAG525 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 29 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
day*ug/mL
  Cycle 1, ROW patients: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 10 | 5 | 6 | 6 | 6 | 5 | 6 | 19 | 4 | 9 | 7 | 3 | 10 | 6 | 11 | 6 | 5
  Cycle 1, ROW patients | 136 (49.2) | 506 (111) | 758 (172) | 1830 (627) | 2810 (555) | 500 (147) | 708 (199) | 631 (184) | 1220 (491) | 2230 (731) | 1290 (537) | 35.8 (10.5) | 174 (31.3) | 138 (38.9) | 162 (56.5) | 588 (196) | 608 (165) | 952 (441) | 1640 (539) | 198 (101) | 1040 (183) | 2890 (982) | 3020 (928) | 150 (61.6) | 484 (173) | 551 (205)
  Cycle 3, ROW patients: number analyzed (Participants) | 4 | 7 | 1 | 1 | 4 | 11 | 9 | 3 | 3 | 2 | 2 | 3 | 5 | 3 | 3 | 4 | 14 | 3 | 6 | 3 | 2 | 4 | 2 | 7 | 4 | 5
  Cycle 3, ROW patients | 264 (146) | 1000 (358) | 2470 | 2330 | 5270 (1250) | 862 (583) | 1390 (759) | 928 (469) | 1200 (754) | 1770 (2230) | 2740 (2680) | 59.9 (39.3) | 286 (134) | 264 (133) | 234 (108) | 1310 (701) | 869 (328) | 1410 (831) | 1990 (1180) | 336 (439) | 2250 (44.7) | 3840 (1600) | 7160 (3190) | 211 (150) | 938 (141) | 1230 (617)
  Cycle 1, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Japanese patients | 144 (35.6) |  |  |  |  | 679 (142) | 1130 (153) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3, Japanese patients: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3, Japanese patients | 89.6 (76.7) |  |  |  |  | 1720 | 2520 (359) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

14. Secondary Outcome: Phase 2: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of LAG525
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 92
day*ug/mL
  Cycle 1, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  Cycle 1, NSCLC patients | 1260 (509) |  | 955 (272)
  Cycle 3, NSCLC patients: number analyzed (Participants) | 16 | 0 | 16
  Cycle 3, NSCLC patients | 1500 (688) |  | 1260 (554)
  Cycle 1, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  Cycle 1, melanoma patients | 1030 (404) |  | 953 (340)
  Cycle 3, melanoma patients: number analyzed (Participants) | 13 | 0 | 16
  Cycle 3, melanoma patients | 1860 (507) |  | 1680 (754)
  Cycle 1, RCC patients: number analyzed (Participants) | 19 | 0 | 17
  Cycle 1, RCC patients | 979 (366) |  | 886 (429)
  Cycle 3, RCC patients: number analyzed (Participants) | 14 | 0 | 13
  Cycle 3, RCC patients | 1420 (678) |  | 1280 (809)
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 41 | 0 | 16
  Cycle 1, mesothelioma patients | 963 (329) |  | 1070 (350)
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 34 | 0 | 16
  Cycle 3, mesothelioma patients | 1400 (732) |  | 1380 (729)
  Cycle 1, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  Cycle 1, TNBC patients | 1180 (379) | 2010 (807) | 1150 (234)
  Cycle 3, TNBC patients: number analyzed (Participants) | 11 | 7 | 9
  Cycle 3, TNBC patients | 1710 (1090) | 2800 (1210) | 1530 (578)

15. Secondary Outcome: Phase 1: Terminal Elimination Half-life (T1/2) of LAG525
Description: Pharmacokinetic (PK) parameters were calculated based on LAG525 serum concentrations by using non-compartmental methods. Elimination half-life (T1/2) values were calculated as 0.693/terminal elimination rate constant.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 29 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
days
  Cycle 1, ROW patients: number analyzed (Participants) | 11 | 12 | 6 | 6 | 6 | 21 | 19 | 5 | 6 | 9 | 5 | 4 | 6 | 6 | 5 | 6 | 18 | 4 | 9 | 7 | 3 | 9 | 6 | 11 | 5 | 5
  Cycle 1, ROW patients | 7.65 (1.94) | 11.1 (4.12) | 9.99 (2.37) | 12 (4.5) | 12.8 (8) | 10.3 (3.5) | 11.5 (6.59) | 13.5 (4.07) | 13.1 (5.38) | 13.9 (5.15) | 13.6 (7.61) | 3.47 (1.4) | 9.15 (3.86) | 6.5 (3.25) | 7.52 (2.5) | 9.5 (2.78) | 11.5 (3.7) | 11.3 (4.94) | 10.2 (3.68) | 7.49 (4.42) | 15.7 (4.23) | 17.9 (7.88) | 14.4 (3.28) | 5.26 (2.43) | 9.12 (2.07) | 9.36 (2.18)
  Cycle 3, ROW patients: number analyzed (Participants) | 3 | 6 | 1 | 1 | 3 | 7 | 8 | 2 | 2 | 1 | 2 | 3 | 5 | 3 | 2 | 1 | 14 | 2 | 5 | 2 | 2 | 3 | 2 | 6 | 4 | 4
  Cycle 3, ROW patients | 11.2 (2.62) | 14.4 (5.82) | 5.94 | 12.2 | 16.5 (2.87) | 12.1 (5.06) | 18 (9.7) | 15 (2.36) | 20.6 (8.51) | 20.8 | 23.4 (14.6) | 6.15 (2.98) | 9.55 (3.95) | 9.17 (4.36) | 13.1 (0.736) | 14.7 | 14.3 (7.02) | 14.5 (1.24) | 13.8 (4.45) | 11.1 (10.9) | 18.3 (3.58) | 15.1 (5.44) | 26.3 (11.9) | 7.32 (4.94) | 10.8 (1.76) | 15.1 (4.54)
  Cycle 1, Japanese patients: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Japanese patients | 13.7 (10.2) |  |  |  |  | 9.42 (2.27) | 13.8 (4.38) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3, Japanese patients: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3, Japanese patients | 5.49 (2.38) |  |  |  |  | 19.4 | 28.1 (18) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

16. Secondary Outcome: Phase 2: Terminal Elimination Half-life (T1/2) of LAG525
Description: as for outcome 15
Time Frame: as for outcome 10
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 and had a valid measure of the endpoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 84 | 13 | 64
days
  Cycle 1, NSCLC patients: number analyzed (Participants) | 17 | 0 | 13
  Cycle 1, NSCLC patients | 11.6 (6.11) |  | 13.3 (4.62)
  Cycle 3, NSCLC patients: number analyzed (Participants) | 9 | 0 | 9
  Cycle 3, NSCLC patients | 16.3 (9.17) |  | 15.9 (7.88)
  Cycle 1, melanoma patients: number analyzed (Participants) | 12 | 0 | 15
  Cycle 1, melanoma patients | 15.6 (5.18) |  | 15.5 (5.92)
  Cycle 3, melanoma patients: number analyzed (Participants) | 9 | 0 | 6
  Cycle 3, melanoma patients | 20.1 (5.24) |  | 19.2 (9.26)
  Cycle 1, RCC patients: number analyzed (Participants) | 13 | 0 | 11
  Cycle 1, RCC patients | 14.2 (3.61) |  | 14.1 (5.39)
  Cycle 3, RCC patients: number analyzed (Participants) | 8 | 0 | 3
  Cycle 3, RCC patients | 14.1 (3.71) |  | 23.1 (6.33)
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 29 | 0 | 11
  Cycle 1, mesothelioma patients | 13 (5.13) |  | 13.7 (5.27)
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 16 | 0 | 8
  Cycle 3, mesothelioma patients | 18.4 (7.16) |  | 18.7 (5.47)
  Cycle 1, TNBC patients: number analyzed (Participants) | 8 | 13 | 7
  Cycle 1, TNBC patients | 22.5 (18.9) | 14.6 (3.82) | 14.4 (5.01)
  Cycle 3, TNBC patients: number analyzed (Participants) | 6 | 0 | 4
  Cycle 3, TNBC patients | 18.7 (9.14) |  | 19 (4.78)

17. Secondary Outcome: Phase 1: Maximum Observed Serum Concentration (Cmax) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
  Japanese patients were not treated with PDR001 and therefore the PK parameters of this study drug are not applicable.
Time Frame: as for outcome 9
Population: All patients in phase 1 who received at least one full or partial dose of PDR001 and who had at least one serum sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
ug/mL
  Cycle 1, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 6 | 5 | 6 | 14 | 4 | 11 | 7 | 4 | 8 | 5 | 9 | 5 | 6
  Cycle 1, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 19.6 (3.59) | 19.6 (2.77) | 17.7 (3.84) | 58.8 (23.2) | 67.9 (20.4) | 76.2 (20) | 61.5 (22.1) | 85.1 (28) | 65 (11.3) | 87.6 (24.5) | 113 (26.8) | 116 (28.1) | 100 (23.1) | 115 (33.2) | 97.9 (17)
  Cycle 3, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 3 | 3 | 8 | 3 | 7 | 2 | 1 | 3 | 2 | 5 | 5 | 3
  Cycle 3, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 30.4 (11.9) | 28.7 (8.4) | 29.7 (9.97) | 89.5 (28.9) | 168 (20.1) | 97.5 (34.4) | 80 (25.1) | 123 (35.6) | 90.8 (51.2) | 142 | 134 (56.7) | 167 (9.9) | 141 (58.2) | 147 (29.8) | 126 (27.2)

18. Secondary Outcome: Phase 2: Maximum Observed Serum Concentration (Cmax) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: as for outcome 10
Population: All patients in phase 2 who received at least one full or partial dose of PDR001 and who had at least one serum sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 92
ug/mL
  Cycle 1, NSCLC patients: number analyzed (Participants) | 20 | 0 | 20
  Cycle 1, NSCLC patients | 102 (33) |  | 68.9 (17.3)
  Cycle 3, NSCLC patients: number analyzed (Participants) | 16 | 0 | 13
  Cycle 3, NSCLC patients | 118 (36.5) |  | 100 (24.2)
  Cycle 1, melanoma patients: number analyzed (Participants) | 19 | 0 | 20
  Cycle 1, melanoma patients | 75.7 (25.2) |  | 71.3 (26.2)
  Cycle 3, melanoma patients: number analyzed (Participants) | 13 | 0 | 14
  Cycle 3, melanoma patients | 117 (29.8) |  | 105 (43.3)
  Cycle 1, RCC patients: number analyzed (Participants) | 18 | 0 | 15
  Cycle 1, RCC patients | 81 (21.3) |  | 67 (25.8)
  Cycle 3, RCC patients: number analyzed (Participants) | 13 | 0 | 13
  Cycle 3, RCC patients | 104 (23.8) |  | 103 (36.1)
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 35 | 0 | 16
  Cycle 1, mesothelioma patients | 70.5 (21.4) |  | 82.7 (39)
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 33 | 0 | 16
  Cycle 3, mesothelioma patients | 96.5 (31.5) |  | 113 (36.8)
  Cycle 1, TNBC patients: number analyzed (Participants) | 20 | 19 | 13
  Cycle 1, TNBC patients | 91.5 (25.1) | 117 (36.7) | 89.8 (14.8)
  Cycle 3, TNBC patients: number analyzed (Participants) | 11 | 5 | 9
  Cycle 3, TNBC patients | 124 (36.5) | 134 (54) | 123 (18.5)

19. Secondary Outcome: Phase 1: Time to Reach Maximum Serum Concentration (Tmax) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
  Japanese patients were not treated with PDR001 and therefore the PK parameters of this study drug are not applicable.
Time Frame: as for outcome 9
Population: as for outcome 17
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
days
  Cycle 1, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 6 | 5 | 6 | 14 | 4 | 11 | 7 | 4 | 8 | 5 | 9 | 5 | 6
  Cycle 1, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 1.5 [1.47 to 1.62] | 1.5 [1.1 to 1.55] | 1.55 [1.42 to 1.63] | 1.63 [1.52 to 1.78] | 1.51 [0.95 to 1.67] | 1.53 [0.467 to 2.42] | 1.75 [1.5 to 2.08] | 1.53 [1.45 to 2.5] | 1.58 [1.5 to 2.02] | 1.5 [1.47 to 1.72] | 1.66 [1.5 to 2.07] | 1.5 [0.583 to 1.58] | 1.5 [1.5 to 1.58] | 1.58 [0.683 to 2.12] | 1.56 [1.47 to 1.68]
  Cycle 3, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 3 | 3 | 8 | 3 | 7 | 2 | 1 | 3 | 2 | 5 | 5 | 3
  Cycle 3, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 1.5 [1.07 to 1.65] | 1.58 [1.57 to 1.68] | 1.55 [1.52 to 1.58] | 1.72 [1.57 to 17.2] | 1.75 [1.58 to 2.08] | 1.5 [0.45 to 1.72] | 1.5 [1.5 to 1.62] | 1.58 [1 to 2.13] | 1.63 [1.58 to 1.67] | 1.8 [1.8 to 1.8] | 1.53 [1.45 to 2.08] | 1.87 [1.57 to 2.17] | 1.55 [1.52 to 1.6] | 1.55 [0.533 to 2.12] | 1.58 [1.52 to 1.68]

20. Secondary Outcome: Phase 2: Time to Reach Maximum Serum Concentration (Tmax) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 10
Population: as for outcome 18
Measure: Median (Full Range); unit: days
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 92
days
  Cycle 1, NSCLC patients: number analyzed (Participants) | 20 | 0 | 20
  Cycle 1, NSCLC patients | 1.57 [1.52 to 3] |  | 1.57 [1 to 2.12]
  Cycle 3, NSCLC patients: number analyzed (Participants) | 16 | 0 | 13
  Cycle 3, NSCLC patients | 1.57 [1.32 to 2.08] |  | 1.58 [1.47 to 2.08]
  Cycle 1, melanoma patients: number analyzed (Participants) | 19 | 0 | 20
  Cycle 1, melanoma patients | 1.55 [0.35 to 3.08] |  | 1.53 [0.567 to 2.5]
  Cycle 3, melanoma patients: number analyzed (Participants) | 13 | 0 | 14
  Cycle 3, melanoma patients | 1.57 [1.08 to 2.08] |  | 1.53 [0.583 to 1.63]
  Cycle 1, RCC patients: number analyzed (Participants) | 18 | 0 | 15
  Cycle 1, RCC patients | 1.58 [1 to 3.08] |  | 1.57 [0.55 to 2]
  Cycle 3, RCC patients: number analyzed (Participants) | 13 | 0 | 13
  Cycle 3, RCC patients | 1.53 [1.5 to 2.08] |  | 1.58 [1.47 to 2]
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 35 | 0 | 16
  Cycle 1, mesothelioma patients | 1.55 [0.483 to 3] |  | 1.54 [0.5 to 2]
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 33 | 0 | 16
  Cycle 3, mesothelioma patients | 1.52 [0.1 to 2.05] |  | 1.5 [0.283 to 2.08]
  Cycle 1, TNBC patients: number analyzed (Participants) | 20 | 19 | 13
  Cycle 1, TNBC patients | 1.58 [0.5 to 3] | 1.57 [1.45 to 2.92] | 1.53 [0.967 to 2.08]
  Cycle 3, TNBC patients: number analyzed (Participants) | 11 | 5 | 9
  Cycle 3, TNBC patients | 1.6 [1.48 to 2.5] | 1.75 [1.6 to 2.43] | 1.65 [1.5 to 2.42]

21. Secondary Outcome: Phase 1: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation.
  Japanese patients were not treated with PDR001 and therefore the PK parameters of this study drug are not applicable.
Time Frame: as for outcome 9
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
day*ug/mL
  Cycle 1, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 18 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
  Cycle 1, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 114 (17) | 141 (45.4) | 134 (25.7) | 437 (177) | 466 (159) | 601 (238) | 537 (163) | 637 (263) | 591 (207) | 789 (319) | 1290 (441) | 1190 (353) | 1080 (412) | 1110 (335) | 950 (264)
  Cycle 3, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 3 | 3 | 4 | 12 | 3 | 7 | 3 | 2 | 4 | 2 | 8 | 5 | 5
  Cycle 3, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 292 (131) | 268 (151) | 289 (196) | 816 (472) | 1340 (673) | 1180 (447) | 1020 (563) | 939 (572) | 1500 (1450) | 1860 (150) | 1950 (645) | 2840 (531) | 1440 (828) | 1510 (874) | 1310 (700)

22. Secondary Outcome: Phase 2: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation.
Time Frame: as for outcome 10
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 92
day*ug/mL
  Cycle 1, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  Cycle 1, NSCLC patients | 853 (347) |  | 629 (197)
  Cycle 3, NSCLC patients: number analyzed (Participants) | 16 | 0 | 17
  Cycle 3, NSCLC patients | 1020 (500) |  | 881 (443)
  Cycle 1, melanoma patients: number analyzed (Participants) | 20 | 0 | 22
  Cycle 1, melanoma patients | 663 (291) |  | 633 (310)
  Cycle 3, melanoma patients: number analyzed (Participants) | 13 | 0 | 16
  Cycle 3, melanoma patients | 1390 (406) |  | 1070 (537)
  Cycle 1, RCC patients: number analyzed (Participants) | 18 | 0 | 17
  Cycle 1, RCC patients | 739 (227) |  | 617 (347)
  Cycle 3, RCC patients: number analyzed (Participants) | 14 | 0 | 14
  Cycle 3, RCC patients | 879 (547) |  | 1060 (464)
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 40 | 0 | 16
  Cycle 1, mesothelioma patients | 633 (263) |  | 747 (388)
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 34 | 0 | 16
  Cycle 3, mesothelioma patients | 1110 (500) |  | 1110 (606)
  Cycle 1, TNBC patients: number analyzed (Participants) | 21 | 21 | 14
  Cycle 1, TNBC patients | 808 (331) | 1110 (621) | 766 (277)
  Cycle 3, TNBC patients: number analyzed (Participants) | 11 | 7 | 9
  Cycle 3, TNBC patients | 1370 (570) | 2150 (1180) | 1360 (351)

23. Secondary Outcome: Phase 1: Terminal Elimination Half-life (T1/2) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Elimination half-life (T1/2) values were calculated as 0.693/terminal elimination rate constant.
  Japanese patients were not treated with PDR001 and therefore the PK parameters of this study drug are not applicable.
Time Frame: as for outcome 9
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 6 | 20 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
day
  Cycle 1, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 6 | 5 | 6 | 16 | 5 | 11 | 7 | 4 | 10 | 6 | 11 | 6 | 6
  Cycle 1, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 9.71 (8.24) | 10.2 (4.81) | 12.5 (3.38) | 20.7 (8.72) | 30.8 (47) | 22.8 (13.8) | 14.8 (4.78) | 11.8 (5) | 14 (3.72) | 15.1 (10.2) | 20.4 (8.41) | 18.7 (7.18) | 20.4 (10) | 14.6 (5.48) | 17.3 (2.76)
  Cycle 3, ROW patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 3 | 2 | 3 | 12 | 3 | 6 | 3 | 1 | 3 | 2 | 7 | 4 | 5
  Cycle 3, ROW patients |  |  |  |  |  |  |  |  |  |  |  | 21.4 (9.4) | 22.3 (7.13) | 12.4 (10.3) | 17.8 (5.03) | 44.4 (36.8) | 27.7 (19.4) | 27.4 (4.25) | 17.4 (5.64) | 20.8 (12.4) | 22.4 | 21.9 (4.22) | 32.8 (12.5) | 16.7 (10.2) | 16.1 (5.64) | 24.9 (6.75)

24. Secondary Outcome: Phase 2: Terminal Elimination Half-life (T1/2) of PDR001
Description: Pharmacokinetic (PK) parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Elimination half-life (T1/2) values were calculated as 0.693/terminal elimination rate constant.
Time Frame: as for outcome 10
Population: All patients in phase 2 who received at least one full or partial dose of PDR001 and had a valid measure of the endpoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 89 | 15 | 61
days
  Cycle 1, NSCLC patients: number analyzed (Participants) | 19 | 0 | 14
  Cycle 1, NSCLC patients | 17.2 (10) |  | 15.8 (5.65)
  Cycle 3, NSCLC patients: number analyzed (Participants) | 7 | 0 | 7
  Cycle 3, NSCLC patients | 16.8 (7.88) |  | 24.5 (8.47)
  Cycle 1, melanoma patients: number analyzed (Participants) | 14 | 0 | 14
  Cycle 1, melanoma patients | 29.1 (31.6) |  | 20 (5.66)
  Cycle 3, melanoma patients: number analyzed (Participants) | 12 | 0 | 10
  Cycle 3, melanoma patients | 24.2 (6.17) |  | 25.6 (15.7)
  Cycle 1, RCC patients: number analyzed (Participants) | 13 | 0 | 9
  Cycle 1, RCC patients | 17.8 (4.77) |  | 18.4 (7.3)
  Cycle 3, RCC patients: number analyzed (Participants) | 10 | 0 | 3
  Cycle 3, RCC patients | 18.4 (5.02) |  | 24.2 (5.05)
  Cycle 1, mesothelioma patients: number analyzed (Participants) | 28 | 0 | 8
  Cycle 1, mesothelioma patients | 19.1 (7.98) |  | 25.6 (7.49)
  Cycle 3, mesothelioma patients: number analyzed (Participants) | 15 | 0 | 7
  Cycle 3, mesothelioma patients | 25.2 (14.5) |  | 17.3 (8.11)
  Cycle 1, TNBC patients: number analyzed (Participants) | 12 | 14 | 8
  Cycle 1, TNBC patients | 18.8 (8.33) | 21.3 (7.43) | 19.9 (6.24)
  Cycle 3, TNBC patients: number analyzed (Participants) | 6 | 2 | 4
  Cycle 3, TNBC patients | 23.9 (17.1) | 22.2 (0.591) | 23.8 (5.64)

25. Secondary Outcome: Phase 1: Number of Participants With Anti-LAG525 Antibodies
Description: Validated immunoassays were used for screening and confirmation of the presence of anti-LAG525 antibodies (ADA, anti-drug antibodies) in serum. Number of participants with ADA in each category is reported in this record.
Time Frame: Baseline (pre-infusion on Cycle 1 Day 1) and post-baseline (assessed throughout the treatment up to maximum 4.4 years).
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 and who had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample. A determinant IG sample is neither ADA-inconclusive nor unevaluable. Japanese patients were analyzed together with the rest of the world (ROW) patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 14 | 11 | 4 | 5 | 6 | 21 | 17 | 4 | 6 | 7 | 5 | 5 | 6 | 5 | 5 | 5 | 15 | 3 | 8 | 6 | 3 | 9 | 5 | 10 | 6 | 5
Participants
  ADA-negative at baseline | 14 | 10 | 4 | 5 | 5 | 19 | 15 | 3 | 6 | 6 | 5 | 5 | 5 | 5 | 4 | 4 | 12 | 3 | 8 | 6 | 3 | 9 | 5 | 10 | 5 | 5
  ADA-positive at post-baseline | 6 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 3 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 5 | 1 | 1

26. Secondary Outcome: Phase 2: Number of Participants With Anti-LAG525 Antibodies
Description: as for outcome 25
Time Frame: Baseline (pre-infusion on Cycle 1 Day 1) and post-baseline (assessed throughout the treatment up to maximum 2.6 years).
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 and who had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample. A determinant IG sample is neither ADA-inconclusive nor unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 106 | 16 | 80
Participants
  ADA-negative at baseline, NSCLC patients: number analyzed (Participants) | 20 | 0 | 20
  ADA-negative at baseline, NSCLC patients | 19 |  | 19
  ADA-positive at post-baseline, NSCLC patients: number analyzed (Participants) | 20 | 0 | 20
  ADA-positive at post-baseline, NSCLC patients | 4 |  | 2
  ADA-negative at baseline, melanoma patients: number analyzed (Participants) | 16 | 0 | 19
  ADA-negative at baseline, melanoma patients | 15 |  | 19
  ADA-positive at post-baseline, melanoma patients: number analyzed (Participants) | 16 | 0 | 19
  ADA-positive at post-baseline, melanoma patients | 1 |  | 0
  ADA-negative at baseline, RCC patients: number analyzed (Participants) | 17 | 0 | 15
  ADA-negative at baseline, RCC patients | 17 |  | 13
  ADA-positive at post-baseline, RCC patients: number analyzed (Participants) | 17 | 0 | 15
  ADA-positive at post-baseline, RCC patients | 0 |  | 1
  ADA-negative at baseline, mesothelioma patients: number analyzed (Participants) | 38 | 0 | 15
  ADA-negative at baseline, mesothelioma patients | 35 |  | 13
  ADA-positive at post-baseline, mesothelioma patients: number analyzed (Participants) | 38 | 0 | 15
  ADA-positive at post-baseline, mesothelioma patients | 3 |  | 1
  ADA-negative at baseline, TNBC patients: number analyzed (Participants) | 15 | 16 | 11
  ADA-negative at baseline, TNBC patients | 15 | 15 | 11
  ADA-positive at post-baseline, TNBC patients: number analyzed (Participants) | 15 | 16 | 11
  ADA-positive at post-baseline, TNBC patients | 2 | 0 | 1

27. Secondary Outcome: Phase 1: Number of Participants With Anti-PDR001 Antibodies
Description: Validated immunoassays were used for screening and confirmation of the presence of anti-PDR001 antibodies (ADA, anti-drug antibodies) in serum. Number of participants with ADA in each category is reported in this record.
Time Frame: Baseline (pre-infusion on Cycle 1 Day 1) and post-baseline (assessed throughout the treatment up to maximum 4.4 years).
Population: All patients in phase 1 who received at least one full or partial dose of PDR001 and who had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample. A determinant IG sample is neither ADA-inconclusive nor unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 5 | 5 | 5 | 16 | 2 | 7 | 7 | 4 | 5 | 2 | 6 | 4 | 3
Participants
  ADA-negative at baseline |  |  |  |  |  |  |  |  |  |  |  | 5 | 6 | 5 | 4 | 5 | 14 | 2 | 7 | 7 | 4 | 5 | 2 | 6 | 3 | 3
  ADA-positive at post-baseline (i.e. ADA incidence) |  |  |  |  |  |  |  |  |  |  |  | 2 | 2 | 2 | 0 | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0

28. Secondary Outcome: Phase 2: Number of Participants With Anti-PDR001 Antibodies
Description: as for outcome 27
Time Frame: Baseline (pre-infusion on Cycle 1 Day 1) and post-baseline (assessed throughout the treatment up to maximum 2.6 years).
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 108 | 14 | 82
Participants
  ADA-negative at baseline, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  ADA-negative at baseline, NSCLC patients | 18 |  | 21
  ADA-positive at post-baseline, NSCLC patients: number analyzed (Participants) | 20 | 0 | 22
  ADA-positive at post-baseline, NSCLC patients | 6 |  | 4
  ADA-negative at baseline, melanoma patients: number analyzed (Participants) | 17 | 0 | 19
  ADA-negative at baseline, melanoma patients | 16 |  | 19
  ADA-positive at post-baseline, melanoma patients: number analyzed (Participants) | 17 | 0 | 19
  ADA-positive at post-baseline, melanoma patients | 5 |  | 0
  ADA-negative at baseline, RCC patients: number analyzed (Participants) | 17 | 0 | 15
  ADA-negative at baseline, RCC patients | 17 |  | 12
  ADA-positive at post-baseline, RCC patients: number analyzed (Participants) | 17 | 0 | 15
  ADA-positive at post-baseline, RCC patients | 2 |  | 0
  ADA-negative at baseline, mesothelioma patients: number analyzed (Participants) | 37 | 0 | 16
  ADA-negative at baseline, mesothelioma patients | 32 |  | 11
  ADA-positive at post-baseline, mesothelioma patients: number analyzed (Participants) | 37 | 0 | 16
  ADA-positive at post-baseline, mesothelioma patients | 6 |  | 2
  ADA-negative at baseline, TNBC patients: number analyzed (Participants) | 17 | 14 | 10
  ADA-negative at baseline, TNBC patients | 17 | 13 | 9
  ADA-positive at post-baseline, TNBC patients: number analyzed (Participants) | 17 | 14 | 10
  ADA-positive at post-baseline, TNBC patients | 5 | 1 | 0

29. Secondary Outcome: Phase 1: Overall Response Rate (ORR) Per RECIST 1.1
Description: Tumor response was based on local investigator assessment and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). ORR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
  ORR is reported for ROW and Japanese patients.
Time Frame: From start of treatment until end of treatment, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
percentage of participants
  ROW: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  ROW | 0 [0.0 to 20.6] | 0 [0.0 to 22.1] | 0 [0.0 to 39.3] | 0 [0.0 to 39.3] | 0 [0.0 to 39.3] | 0 [0.0 to 11.3] | 0 [0.0 to 11.7] | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] | 0 [0.0 to 23.8] | 0 [0.0 to 45.1] | 33.3 [6.3 to 72.9] | 0 [0.0 to 39.3] | 16.7 [0.9 to 58.2] | 0 [0.0 to 45.1] | 16.7 [0.9 to 58.2] | 20.0 [7.1 to 40.1] | 33.3 [6.3 to 72.9] | 0 [0.0 to 22.1] | 0 [0.0 to 34.8] | 0 [0.0 to 39.3] | 16.7 [3.0 to 43.8] | 0 [0.0 to 39.3] | 0 [0.0 to 23.8] | 16.7 [0.9 to 58.2] | 0 [0.0 to 39.3]
  Japanese: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 0 [0.0 to 52.7] |  |  |  |  | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

30. Secondary Outcome: Phase 1: Overall Response Rate (ORR) Per irRC
Description: TTumor response was based on local investigator assessment and the assessment criteria was immune-related Response Criteria (irRC). ORR per irRC is defined as the percentage of participants with a best overall response of immune related Complete Response (irCR) or immune related Partial Response (irPR).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new target lesions, taking as reference the baseline sum of diameters.
  ORR is reported for ROW and Japanese patients.
Time Frame: From start of treatment until end of treatment, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
percentage of participants
  ROW: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  ROW | 0 [0.0 to 20.6] | 0 [0.0 to 22.1] | 0 [0.0 to 39.3] | 0 [0.0 to 39.3] | 0 [0.0 to 39.3] | 0 [0.0 to 11.3] | 0 [0.0 to 11.7] | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] | 0 [0.0 to 23.8] | 0 [0.0 to 45.1] | 33.3 [6.3 to 72.9] | 0 [0.0 to 39.3] | 16.7 [0.9 to 58.2] | 0 [0.0 to 45.1] | 16.7 [0.9 to 58.2] | 20.0 [7.1 to 40.1] | 33.3 [6.3 to 72.9] | 0 [0.0 to 22.1] | 0 [0.0 to 34.8] | 0 [0.0 to 39.3] | 33.3 [12.3 to 60.9] | 0 [0.0 to 39.3] | 0 [0.0 to 23.8] | 16.7 [0.9 to 58.2] | 0 [0.0 to 39.3]
  Japanese: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 0 [0.0 to 52.7] |  |  |  |  | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

31. Secondary Outcome: Phase 2: Overall Response Rate (ORR) Per irRC
Description: Tumor response was based on local investigator assessment and the assessment criteria was immune-related Response Criteria (irRC). ORR per irRC is defined as the percentage of participants with a best overall response of immune related Complete Response (irCR) or immune related Partial Response (irPR).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new target lesions, taking as reference the baseline sum of diameters.
  ORR is reported by tumor type.
Time Frame: From start of treatment until end of treatment, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
percentage of participants
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  Non-small cell lung cancer (NSCLC) | 15.0 [4.2 to 34.4] |  | 0 [0.0 to 12.7]
  Melanoma: number analyzed (Participants) | 20 | 0 | 22
  Melanoma | 15.0 [4.2 to 34.4] |  | 9.1 [1.6 to 25.9]
  Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  Renal cell cancer (RCC) | 26.3 [11.0 to 47.6] |  | 5.3 [0.3 to 22.6]
  Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  Mesothelioma | 19.5 [10.1 to 32.5] |  | 6.3 [0.3 to 26.4]
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  Triple negative breast cancer (TNBC) | 14.3 [4.0 to 32.9] | 4.8 [0.2 to 20.7] | 0 [0.0 to 19.3]

32. Secondary Outcome: Phase 1: Disease Control Rate (DCR) Per RECIST 1.1
Description: Tumor response was based on local investigator assessment and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). DCR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
  DCR is reported for ROW and Japanese patients.
Time Frame: From start of treatment until end of treatment, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
percentage of participants
  ROW: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  ROW | 23.1 [6.6 to 49.5] | 41.7 [18.1 to 68.5] | 16.7 [0.9 to 58.2] | 0 [0.0 to 39.3] | 66.7 [27.1 to 93.7] | 24.0 [11.0 to 42.0] | 20.8 [8.6 to 38.9] | 20.0 [1.0 to 65.7] | 33.3 [6.3 to 72.9] | 18.2 [3.3 to 47.0] | 20.0 [1.0 to 65.7] | 50.0 [15.3 to 84.7] | 33.3 [6.3 to 72.9] | 33.3 [6.3 to 72.9] | 60.0 [18.9 to 92.4] | 33.3 [6.3 to 72.9] | 55.0 [34.7 to 74.1] | 50.0 [15.3 to 84.7] | 8.3 [0.4 to 33.9] | 28.6 [5.3 to 65.9] | 66.7 [27.1 to 93.7] | 41.7 [18.1 to 68.5] | 16.7 [0.9 to 58.2] | 36.4 [13.5 to 65.0] | 50.0 [15.3 to 84.7] | 50.0 [15.3 to 84.7]
  Japanese: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 25.0 [1.3 to 75.1] |  |  |  |  | 40.0 [7.6 to 81.1] | 16.7 [0.9 to 58.2] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

33. Secondary Outcome: Phase 1: Disease Control Rate (DCR) Per irRC
Description: Tumor response was based on local investigator assessment and the assessment criteria was immune-related Response Criteria (irRC). DCR per irRC is defined as the percentage of participants with a best overall response of immune related Complete Response (irCR), immune related Partial Response (irPR) or immune related Stable Disease (irSD).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for irPR or irCR nor an increase in lesions which would qualify for progression.
  DCR is reported for ROW and Japanese patients.
Time Frame: From start of treatment until end of treatment, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
percentage of participants
  ROW: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  ROW | 30.8 [11.3 to 57.3] | 33.3 [12.3 to 60.9] | 16.7 [0.9 to 58.2] | 0 [0.0 to 39.3] | 50.0 [15.3 to 84.7] | 28.0 [13.9 to 46.2] | 33.3 [17.8 to 52.1] | 20.0 [1.0 to 65.7] | 33.3 [6.3 to 72.9] | 18.2 [3.3 to 47.0] | 20.0 [1.0 to 65.7] | 50.0 [15.3 to 84.7] | 66.7 [27.1 to 93.7] | 50.0 [15.3 to 84.7] | 60.0 [18.9 to 92.4] | 33.3 [6.3 to 72.9] | 55.0 [34.7 to 74.1] | 50.0 [15.3 to 84.7] | 8.3 [0.4 to 33.9] | 28.6 [5.3 to 65.9] | 66.7 [27.1 to 93.7] | 50.0 [24.5 to 75.5] | 33.3 [6.3 to 72.9] | 36.4 [13.5 to 65.0] | 50.0 [15.3 to 84.7] | 50.0 [15.3 to 84.7]
  Japanese: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 25.0 [1.3 to 75.1] |  |  |  |  | 40.0 [7.6 to 81.1] | 16.7 [0.9 to 58.2] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

34. Secondary Outcome: Phase 2: Disease Control Rate (DCR) Per RECIST 1.1
Description: Tumor response was based on local investigator assessment and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). DCR per RECIST 1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
  DCR is reported by tumor type.
Time Frame: From start of treatment until end of treatment, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
percentage of participants
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  Non-small cell lung cancer (NSCLC) | 50.0 [30.2 to 69.8] |  | 50.0 [31.1 to 68.9]
  Melanoma: number analyzed (Participants) | 20 | 0 | 22
  Melanoma | 45.0 [25.9 to 65.3] |  | 40.9 [23.3 to 60.5]
  Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  Renal cell cancer (RCC) | 63.2 [41.8 to 81.2] |  | 42.1 [23.0 to 63.2]
  Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  Mesothelioma | 65.9 [51.9 to 78.0] |  | 56.3 [33.3 to 77.3]
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  Triple negative breast cancer (TNBC) | 33.3 [16.8 to 53.6] | 23.8 [9.9 to 43.7] | 21.4 [6.1 to 46.6]

35. Secondary Outcome: Phase 2: Disease Control Rate (DCR) Per irRC
Description: Tumor response was based on local investigator assessment and the assessment criteria was immune-related Response Criteria (irRC). DCR per irRC is defined as the percentage of participants with a best overall response of immune related Complete Response (irCR), immune related Partial Response (irPR) or immune related Stable Disease (irSD).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for irPR or irCR nor an increase in lesions which would qualify for progression.
  DCR is reported by tumor type.
Time Frame: From start of treatment until end of treatment, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
percentage of participants
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  Non-small cell lung cancer (NSCLC) | 60.0 [39.4 to 78.3] |  | 50.0 [31.1 to 68.9]
  Melanoma: number analyzed (Participants) | 20 | 0 | 22
  Melanoma | 55.0 [34.7 to 74.1] |  | 40.9 [23.3 to 60.5]
  Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  Renal cell cancer (RCC) | 68.4 [47.0 to 85.3] |  | 42.1 [23.0 to 63.2]
  Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  Mesothelioma | 65.9 [51.9 to 78.0] |  | 56.3 [33.3 to 77.3]
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  Triple negative breast cancer (TNBC) | 33.3 [16.8 to 53.6] | 28.6 [13.2 to 48.7] | 21.4 [6.1 to 46.6]

36. Secondary Outcome: Phase 1: Duration of Response (DOR) Per RECIST 1.1
Description: DOR only applies to subjects for whom best overall response is complete response (CR) or partial response (PR). DOR is defined as the time from the date of first documented response (CR or PR) to the date of first documented progression or death due to study indication. If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was RECIST 1.1.
Time Frame: From first documented response (CR or PR) to first documented progression or death due to study indication, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001 and had a documented response (CR or PR).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
months |  |  |  |  |  |  |  |  |  |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | 12.2 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [7.9 to NA] — Not estimable due to insufficient number of participants with events. | 18.4 [2.8 to NA] — Not estimable due to insufficient number of participants with events. |  |  |  | 6.5 [5.6 to NA] — Not estimable due to insufficient number of participants with events. |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |

37. Secondary Outcome: Phase 1: Duration of Response (DOR) Per irRC
Description: DOR only applies to subjects for whom best overall response is immune related complete response (irCR) or immune related partial response (irPR). DOR is defined as the time from the date of first documented response (irCR or irPR) to the date of first documented progression or death due to study indication. If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was irRC.
Time Frame: From first documented response (irCR or irPR) to first documented progression or death due to study indication, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001 and had a documented response (irCR or irPR).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
months |  |  |  |  |  |  |  |  |  |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  | 12.2 [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [7.9 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  |  |  | 9.2 [4.4 to NA] — Not estimable due to insufficient number of participants with events. |  |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |

38. Secondary Outcome: Phase 2: Duration of Response (DOR) Per RECIST 1.1
Description: DOR only applies to subjects for whom best overall response is complete response (CR) or partial response (PR). DOR is defined as the time from the date of first documented response (CR or PR) to the date of first documented progression or death due to study indication. If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was RECIST 1.1.
  DOR is reported by tumor type.
Time Frame: From first documented response (CR or PR) to first documented progression or death due to study indication, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001 and had a documented response (CR or PR).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 21 | 1 | 4
months
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 3 | 0 | 0
  Non-small cell lung cancer (NSCLC) | 5.0 [3.7 to NA] — Not estimable due to insufficient number of participants with events. |  |
  Melanoma: number analyzed (Participants) | 3 | 0 | 2
  Melanoma | 11.0 [4.2 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [18.2 to NA] — Not estimable due to insufficient number of participants with events.
  Renal cell cancer (RCC): number analyzed (Participants) | 5 | 0 | 1
  Renal cell cancer (RCC) | NA [7.6 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events.
  Mesothelioma: number analyzed (Participants) | 7 | 0 | 1
  Mesothelioma | NA [5.8 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events.
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 3 | 1 | 0
  Triple negative breast cancer (TNBC) | NA [7.6 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |

39. Secondary Outcome: Phase 2: Duration of Response (DOR) Per irRC
Description: DOR only applies to subjects for whom best overall response is immune related complete response (irCR) or immune related partial response (irPR). DOR is defined as the time from the date of first documented response (irCR or irPR) to the date of first documented progression or death due to study indication. If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was irRC.
  DOR is reported by tumor type.
Time Frame: From first documented response (irCR or irPR) to first documented progression or death due to study indication, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001 and had a documented response (irCR or irPR).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 22 | 1 | 4
months
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 3 | 0 | 0
  Non-small cell lung cancer (NSCLC) | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |  |
  Melanoma: number analyzed (Participants) | 3 | 0 | 2
  Melanoma | 17.5 [11.0 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [18.2 to NA] — Not estimable due to insufficient number of participants with events.
  Renal cell cancer (RCC): number analyzed (Participants) | 5 | 0 | 1
  Renal cell cancer (RCC) | NA [7.6 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events.
  Mesothelioma: number analyzed (Participants) | 8 | 0 | 1
  Mesothelioma | NA [5.8 to NA] — Not estimable due to insufficient number of participants with events. |  | NA [NA to NA] — Not estimable due to insufficient number of participants with events.
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 3 | 1 | 0
  Triple negative breast cancer (TNBC) | NA [7.6 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events. |

40. Secondary Outcome: Phase 1: Progression-free Survival (PFS) Per RECIST 1.1
Description: PFS is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was RECIST 1.1.
  PFS is reported for ROW and Japanese patients.
Time Frame: From start of treatment to first documented progression or death due to any cause, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
months
  ROW: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  ROW | 1.8 [1.6 to 2.0] | 2.3 [1.7 to 3.5] | 1.6 [0.8 to 1.9] | 1.9 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 7.9 [1.3 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [1.6 to 1.9] | 1.8 [1.5 to 1.9] | 2.8 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 2.1 [0.3 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.0 to 2.0] | 1.5 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 3.8 [1.3 to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.8 to 3.5] | 1.8 [1.1 to 3.4] | 8.4 [1.7 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 2.8 [2.0 to 4.2] | 6.5 [0.6 to NA] — Not estimable due to insufficient number of participants with events. | 1.4 [0.6 to 1.8] | 1.8 [1.2 to 2.5] | 3.1 [1.0 to 5.0] | 2.3 [1.6 to 5.7] | 1.5 [0.9 to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.7 to 2.9] | 3.8 [1.6 to 7.6] | 3.2 [1.7 to 5.8]
  Japanese: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 1.8 [1.2 to NA] — Not estimable due to insufficient number of participants with events. |  |  |  |  | 1.8 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [1.2 to 1.8] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

41. Secondary Outcome: Phase 1: Progression-free Survival (PFS) Per irRC
Description: PFS is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was irRC.
  PFS is reported for ROW and Japanese patients.
Time Frame: From start of treatment to first documented progression or death due to any cause, assessed up to 4.4 years
Population: All patients in phase 1 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W
Number analyzed (Participants) | 17 | 12 | 6 | 6 | 6 | 30 | 30 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
months
  ROW: number analyzed (Participants) | 13 | 12 | 6 | 6 | 6 | 25 | 24 | 5 | 6 | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 20 | 6 | 12 | 7 | 6 | 12 | 6 | 11 | 6 | 6
  ROW | 1.9 [1.6 to 2.7] | 1.9 [1.7 to 3.4] | 1.6 [0.8 to 1.9] | 1.9 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 3.4 [1.3 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.6 to 1.9] | 1.9 [1.5 to 2.3] | 2.8 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 2.6 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.0 to 2.0] | 1.5 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 3.8 [1.3 to NA] — Not estimable due to insufficient number of participants with events. | 4.2 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 2.6 [1.1 to NA] — Not estimable due to insufficient number of participants with events. | 8.4 [1.7 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 2.8 [2.0 to 4.2] | 7.5 [0.6 to NA] — Not estimable due to insufficient number of participants with events. | 1.6 [0.6 to 1.8] | 2.0 [1.5 to 2.5] | 3.1 [1.0 to 5.0] | 3.2 [1.7 to 9.1] | 1.5 [0.9 to NA] — Not estimable due to insufficient number of participants with events. | 2.0 [1.7 to 4.2] | 3.8 [1.6 to 7.6] | 3.2 [1.7 to 5.8]
  Japanese: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese | 1.8 [1.2 to NA] — Not estimable due to insufficient number of participants with events. |  |  |  |  | 1.8 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [1.2 to 1.8] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

42. Secondary Outcome: Phase 2: Progression-free Survival (PFS) Per RECIST 1.1
Description: PFS is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was RECIST 1.1.
  PFS is reported by tumor type.
Time Frame: From start of treatment to first documented progression or death due to any cause, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
months
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  Non-small cell lung cancer (NSCLC) | 3.9 [1.7 to 5.6] |  | 3.5 [1.9 to 4.9]
  Melanoma: number analyzed (Participants) | 20 | 0 | 22
  Melanoma | 2.2 [1.6 to 5.6] |  | 1.9 [1.8 to 3.7]
  Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  Renal cell cancer (RCC) | 4.4 [2.1 to 11.1] |  | 3.0 [1.6 to 3.9]
  Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  Mesothelioma | 5.5 [3.5 to 6.4] |  | 3.4 [1.8 to 3.8]
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  Triple negative breast cancer (TNBC) | 1.9 [1.5 to 3.5] | 1.8 [1.4 to 2.6] | 1.7 [1.3 to 3.4]

43. Secondary Outcome: Phase 2: Progression-free Survival (PFS) Per irRC
Description: PFS is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
  Tumor response was based on local investigator assessment and the assessment criteria was irRC.
  PFS is reported by tumor type.
Time Frame: From start of treatment to first documented progression or death due to any cause, assessed up to 2.6 years
Population: All patients in phase 2 who received at least one full or partial dose of LAG525 or PDR001.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: Naive - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated - LAG525 400 mg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 121 | 21 | 93
months
  Non-small cell lung cancer (NSCLC): number analyzed (Participants) | 20 | 0 | 22
  Non-small cell lung cancer (NSCLC) | 4.2 [1.7 to 7.4] |  | 3.5 [1.9 to 4.9]
  Melanoma: number analyzed (Participants) | 20 | 0 | 22
  Melanoma | 5.4 [1.6 to 5.6] |  | 1.9 [1.8 to 3.7]
  Renal cell cancer (RCC): number analyzed (Participants) | 19 | 0 | 19
  Renal cell cancer (RCC) | 5.8 [4.4 to 11.1] |  | 3.0 [1.6 to 3.9]
  Mesothelioma: number analyzed (Participants) | 41 | 0 | 16
  Mesothelioma | 5.6 [3.5 to 7.4] |  | 3.4 [1.8 to 5.7]
  Triple negative breast cancer (TNBC): number analyzed (Participants) | 21 | 21 | 14
  Triple negative breast cancer (TNBC) | 1.9 [1.5 to 3.8] | 1.9 [1.4 to 3.6] | 1.7 [1.3 to 3.4]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until last dose of study treatment plus 30 days, up to maximum 4.5 years (phase 1) and 2.7 years (phase 2).
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment.
Groups:
- Phase 1: LAG525 1 mg/kg Q2W: Single-agent LAG525 1 mg/kg Q2W (ROW patients)
- Phase 1: LAG525 240 mg Q2W: Single-agent LAG525 240 mg Q2W (ROW patients)
- Phase 1: LAG525 400 mg Q2W: Single-agent LAG525 400 mg Q2W (ROW patients)
- Phase 1: LAG525 1 mg/kg Q2W-JP: Single-agent LAG525 1 mg/kg Q2W (Japanese patients)
- Phase 1: LAG525 240 mg Q2W-JP: Single-agent LAG525 240 mg Q2W (Japanese patients)
- Phase 1: LAG525 400 mg Q2W-JP: Single-agent LAG525 400 mg Q2W (Japanese patients)
- Phase 2: Naive - NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with NSCLC naïve to anti-PD-1/PD-L1
- Phase 2: Naive - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with melanoma naïve to anti-PD-1/PD-L1
- Phase 2: Naive - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with RCC naïve to anti-PD-1/PD-L1
- Phase 2: Naive - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with mesothelioma naïve to anti-PD-1/PD-L1
- Phase 2: Naive - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with TNBC naïve to anti-PD-1/PD-L1
- Phase 2: Naive - TNBC - LAG525 600 mg Q4W + PDR001 400 mg Q4W: Combination LAG525 600 mg + PDR001 400 mg (Q4W/Q4W) in patients with TNBC naïve to anti-PD-1/PD-L1
- Phase 2: Pre-treated -NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with NSCLC pre-treated with anti-PD-1/PD-L1
- Phase 2: Pre-treated - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with melanoma pre-treated with anti-PD-1/PD-L1
- Phase 2: Pre-treated - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with RCC pre-treated with anti-PD-1/PD-L1
- Phase 2: Pre-treated - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with mesothelioma pre-treated with anti-PD-1/PD-L1
- Phase 2: Pre-treated - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W: Combination LAG525 400 mg + PDR001 300 mg (Q3W/Q3W) in patients with TNBC pre-treated with anti-PD-1/PD-L1
- All Patients: All patients
Arm/Group | Phase 1: LAG525 1 mg/kg Q2W | Phase 1: LAG525 3 mg/kg Q2W | Phase 1: LAG525 5 mg/kg Q2W | Phase 1: LAG525 10 mg/kg Q2W | Phase 1: LAG525 15 mg/kg Q2W | Phase 1: LAG525 240 mg Q2W | Phase 1: LAG525 400 mg Q2W | Phase 1: LAG525 1 mg/kg Q2W-JP | Phase 1: LAG525 240 mg Q2W-JP | Phase 1: LAG525 400 mg Q2W-JP | Phase 1: LAG525 3 mg/kg Q4W | Phase 1: LAG525 5 mg/kg Q4W | Phase 1: LAG525 10 mg/kg Q4W | Phase 1: LAG525 400 mg Q4W | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W | Phase 2: Naive - NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Naive - TNBC - LAG525 600 mg Q4W + PDR001 400 mg Q4W | Phase 2: Pre-treated -NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Pre-treated - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Pre-treated - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Pre-treated - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W | Phase 2: Pre-treated - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W | All Patients
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/12 | 0/6 | 0/6 | 0/6 | 5/25 | 3/24 | 0/4 | 0/5 | 0/6 | 0/5 | 0/6 | 1/11 | 0/5 | 0/6 | 0/6 | 1/6 | 1/5 | 0/6 | 1/20 | 0/6 | 2/12 | 1/7 | 0/6 | 1/12 | 0/6 | 0/11 | 1/6 | 1/6 | 1/20 | 3/20 | 2/19 | 1/41 | 1/21 | 1/21 | 1/22 | 1/22 | 0/19 | 2/16 | 1/14 | 33/490
Serious Adverse Events (participants affected / at risk) | 4/13 | 2/12 | 5/6 | 2/6 | 3/6 | 10/25 | 11/24 | 0/4 | 2/5 | 0/6 | 2/5 | 4/6 | 5/11 | 2/5 | 3/6 | 2/6 | 3/6 | 3/5 | 1/6 | 9/20 | 3/6 | 6/12 | 4/7 | 5/6 | 5/12 | 2/6 | 5/11 | 4/6 | 4/6 | 13/20 | 8/20 | 14/19 | 15/41 | 9/21 | 10/21 | 7/22 | 8/22 | 5/19 | 4/16 | 4/14 | 208/490
Other Adverse Events (participants affected / at risk) | 13/13 | 11/12 | 6/6 | 6/6 | 6/6 | 24/25 | 24/24 | 4/4 | 5/5 | 6/6 | 5/5 | 6/6 | 11/11 | 5/5 | 6/6 | 6/6 | 6/6 | 5/5 | 6/6 | 19/20 | 5/6 | 12/12 | 7/7 | 6/6 | 12/12 | 6/6 | 11/11 | 6/6 | 6/6 | 19/20 | 17/20 | 19/19 | 41/41 | 21/21 | 21/21 | 21/22 | 22/22 | 19/19 | 16/16 | 14/14 | 481/490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: LAG525 1 mg/kg Q2W (N=13) | Phase 1: LAG525 3 mg/kg Q2W (N=12) | Phase 1: LAG525 5 mg/kg Q2W (N=6) | Phase 1: LAG525 10 mg/kg Q2W (N=6) | Phase 1: LAG525 15 mg/kg Q2W (N=6) | Phase 1: LAG525 240 mg Q2W (N=25) | Phase 1: LAG525 400 mg Q2W (N=24) | Phase 1: LAG525 1 mg/kg Q2W-JP (N=4) | Phase 1: LAG525 240 mg Q2W-JP (N=5) | Phase 1: LAG525 400 mg Q2W-JP (N=6) | Phase 1: LAG525 3 mg/kg Q4W (N=5) | Phase 1: LAG525 5 mg/kg Q4W (N=6) | Phase 1: LAG525 10 mg/kg Q4W (N=11) | Phase 1: LAG525 400 mg Q4W (N=5) | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W (N=6) | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W (N=6) | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W (N=6) | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W (N=5) | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W (N=6) | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W (N=20) | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=6) | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W (N=12) | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W (N=7) | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W (N=6) | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W (N=12) | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W (N=6) | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W (N=11) | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W (N=6) | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W (N=6) | Phase 2: Naive - NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=20) | Phase 2: Naive - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=20) | Phase 2: Naive - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=19) | Phase 2: Naive - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=41) | Phase 2: Naive - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=21) | Phase 2: Naive - TNBC - LAG525 600 mg Q4W + PDR001 400 mg Q4W (N=21) | Phase 2: Pre-treated -NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=22) | Phase 2: Pre-treated - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=22) | Phase 2: Pre-treated - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=19) | Phase 2: Pre-treated - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=16) | Phase 2: Pre-treated - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=14) | All Patients (N=490)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 9
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 13
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 8
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 2 | 0 | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 12
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: LAG525 1 mg/kg Q2W (N=13) | Phase 1: LAG525 3 mg/kg Q2W (N=12) | Phase 1: LAG525 5 mg/kg Q2W (N=6) | Phase 1: LAG525 10 mg/kg Q2W (N=6) | Phase 1: LAG525 15 mg/kg Q2W (N=6) | Phase 1: LAG525 240 mg Q2W (N=25) | Phase 1: LAG525 400 mg Q2W (N=24) | Phase 1: LAG525 1 mg/kg Q2W-JP (N=4) | Phase 1: LAG525 240 mg Q2W-JP (N=5) | Phase 1: LAG525 400 mg Q2W-JP (N=6) | Phase 1: LAG525 3 mg/kg Q4W (N=5) | Phase 1: LAG525 5 mg/kg Q4W (N=6) | Phase 1: LAG525 10 mg/kg Q4W (N=11) | Phase 1: LAG525 400 mg Q4W (N=5) | Phase 1: LAG525 0.3 mg/kg Q2W + PDR001 1 mg/kg Q2W (N=6) | Phase 1: LAG525 1 mg/kg Q2W + PDR001 1 mg/kg Q2W (N=6) | Phase 1: LAG525 80 mg Q2W + PDR001 80 mg Q2W (N=6) | Phase 1: LAG525 80 mg Q2W + PDR001 240 mg Q2W (N=5) | Phase 1: LAG525 240 mg Q2W + PDR001 240 mg Q2W (N=6) | Phase 1: LAG525 240 mg Q3W + PDR001 300 mg Q3W (N=20) | Phase 1: LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=6) | Phase 1: LAG525 600 mg Q3W + PDR001 300 mg Q3W (N=12) | Phase 1: LAG525 80 mg Q4W + PDR001 240 mg Q4W (N=7) | Phase 1: LAG525 400 mg Q4W + PDR001 400 mg Q4W (N=6) | Phase 1: LAG525 800 mg Q4W + PDR001 400 mg Q4W (N=12) | Phase 1: LAG525 1000 mg Q4W + PDR001 400 mg Q4W (N=6) | Phase 1: LAG525 80 mg Q2W + PDR001 400 mg Q4W (N=11) | Phase 1: LAG525 240 mg Q2W + PDR001 400 mg Q4W (N=6) | Phase 1: LAG525 300 mg Q2W + PDR001 400 mg Q4W (N=6) | Phase 2: Naive - NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=20) | Phase 2: Naive - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=20) | Phase 2: Naive - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=19) | Phase 2: Naive - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=41) | Phase 2: Naive - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=21) | Phase 2: Naive - TNBC - LAG525 600 mg Q4W + PDR001 400 mg Q4W (N=21) | Phase 2: Pre-treated -NSCLC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=22) | Phase 2: Pre-treated - Melanoma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=22) | Phase 2: Pre-treated - RCC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=19) | Phase 2: Pre-treated - Mesothelioma - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=16) | Phase 2: Pre-treated - TNBC - LAG525 400 mg Q3W + PDR001 300 mg Q3W (N=14) | All Patients (N=490)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 2 | 2 | 3 | 6 | 2 | 3 | 0 | 1 | 3 | 3 | 0 | 2 | 1 | 1 | 1 | 0 | 5 | 1 | 2 | 2 | 2 | 2 | 1 | 4 | 1 | 1 | 2 | 2 | 9 | 3 | 2 | 3 | 1 | 6 | 4 | 1 | 0 | 92
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 11
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 5
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 8
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
External ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 16
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 4 | 5 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 36
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lacrimal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 1 | 14
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 27
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1 | 3 | 6 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 5 | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 1 | 1 | 2 | 6 | 2 | 3 | 1 | 68
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 24
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 13
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 4 | 3 | 6 | 1 | 1 | 2 | 1 | 1 | 4 | 1 | 2 | 0 | 2 | 2 | 0 | 7 | 0 | 2 | 1 | 3 | 3 | 2 | 3 | 0 | 1 | 10 | 4 | 4 | 7 | 2 | 4 | 3 | 4 | 5 | 0 | 0 | 102
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 5 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 10 | 2 | 3 | 0 | 1 | 6 | 2 | 3 | 0 | 4 | 5 | 4 | 4 | 8 | 3 | 2 | 5 | 4 | 1 | 4 | 2 | 91
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 28
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 16
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 11
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 25
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 7
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 1 | 8 | 7 | 0 | 2 | 2 | 0 | 2 | 3 | 1 | 1 | 1 | 2 | 2 | 0 | 9 | 2 | 4 | 3 | 0 | 7 | 1 | 5 | 2 | 3 | 2 | 6 | 5 | 12 | 3 | 5 | 7 | 9 | 3 | 6 | 1 | 134
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 22
Tongue discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 5 | 5 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 1 | 3 | 2 | 4 | 1 | 0 | 4 | 0 | 4 | 1 | 2 | 2 | 1 | 5 | 5 | 3 | 5 | 6 | 4 | 2 | 1 | 1 | 85
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 3 | 0 | 1 | 1 | 9 | 1 | 3 | 5 | 3 | 3 | 1 | 2 | 63
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 10
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Fatigue (General disorders) | 1 | 3 | 2 | 2 | 3 | 7 | 8 | 0 | 0 | 0 | 3 | 1 | 4 | 0 | 2 | 2 | 2 | 3 | 2 | 10 | 1 | 5 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 3 | 9 | 4 | 6 | 2 | 4 | 6 | 8 | 3 | 127
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 9
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Mucosal disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 6 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 29
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 3 | 0 | 3 | 3 | 2 | 1 | 3 | 4 | 2 | 0 | 2 | 2 | 1 | 1 | 2 | 0 | 47
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 23
Peripheral swelling (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 11
Pyrexia (General disorders) | 3 | 0 | 0 | 0 | 1 | 7 | 5 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 2 | 2 | 1 | 2 | 3 | 1 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 4 | 3 | 4 | 7 | 5 | 5 | 4 | 2 | 5 | 2 | 1 | 85
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 4
Erythema migrans (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 14
Infusion site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 8
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 8
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 5
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 16
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 6 | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 25
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 18
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 9
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 34
Amylase increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 24
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 3 | 0 | 3 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 40
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 29
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 17
Blood calcium (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 26
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood prolactin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Blood thyroid stimulating hormone abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Computerised tomogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Hepatitis C virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 2 | 2 | 27
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 13
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Protein urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thyroxine free abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 4 | 3 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 30
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 9
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 2 | 0 | 2 | 6 | 6 | 0 | 3 | 2 | 1 | 0 | 1 | 3 | 3 | 0 | 0 | 2 | 0 | 9 | 0 | 6 | 1 | 3 | 3 | 2 | 3 | 2 | 2 | 4 | 2 | 4 | 11 | 4 | 2 | 6 | 5 | 3 | 3 | 1 | 113
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 3 | 22
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 22
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 25
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 5 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 31
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 28
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 1 | 4 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 4 | 1 | 2 | 1 | 0 | 4 | 2 | 2 | 1 | 1 | 7 | 4 | 5 | 8 | 6 | 3 | 4 | 7 | 1 | 4 | 1 | 88
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2 | 2 | 4 | 0 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 3 | 2 | 4 | 2 | 0 | 3 | 1 | 3 | 6 | 1 | 2 | 4 | 5 | 1 | 3 | 1 | 69
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 13
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 10
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 9
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 20
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 1 | 3 | 0 | 3 | 0 | 1 | 2 | 1 | 36
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 4 | 1 | 2 | 2 | 2 | 0 | 2 | 0 | 34
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 6
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 11
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Clonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 4 | 0 | 1 | 0 | 2 | 0 | 28
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 15
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 3 | 2 | 2 | 2 | 6 | 5 | 3 | 2 | 56
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 8
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 21
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 7
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 2 | 2 | 36
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 10
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 8
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 10
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Adnexa uteri pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 5
Penile erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 2 | 3 | 5 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 4 | 1 | 1 | 1 | 3 | 3 | 1 | 2 | 0 | 3 | 3 | 1 | 3 | 1 | 0 | 3 | 3 | 5 | 11 | 3 | 4 | 3 | 3 | 5 | 3 | 3 | 94
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1 | 2 | 4 | 7 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 2 | 1 | 3 | 1 | 1 | 6 | 1 | 1 | 0 | 2 | 1 | 1 | 4 | 1 | 0 | 4 | 3 | 5 | 7 | 2 | 5 | 3 | 2 | 2 | 8 | 3 | 95
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 17
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 10
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 16
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 16
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 20
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 12
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 24
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 9
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 7
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 4 | 2 | 3 | 8 | 7 | 5 | 1 | 3 | 1 | 4 | 3 | 64
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 5 | 5 | 7 | 2 | 1 | 1 | 4 | 5 | 3 | 4 | 0 | 57
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 24
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 6
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 8
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 5 | 0 | 2 | 2 | 0 | 0 | 0 | 34
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 22
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 7
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT02460224/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT02460224/SAP_001.pdf